CLINICAL TRIAL: NCT01210768
Title: A Phase II Randomized Study of Pegylated Liposomal Doxorubicin, Cyclophosphamide Versus Epirubicin-Cyclophosphamide as Adjuvant Chemotherapy in Her2-negative Stage I and II Breast Cancer Patients
Brief Title: A Study of Pegylated Liposomal Doxorubicin and Cyclophosphamide in Her2-negative Stage I and II Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTYLD0914
Record Dates: First submitted 2010-08-31; First posted 2010-09-28 (Estimated); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Phase II; Pegylated Liposomal Doxorubicin; Adjuvant Chemotherapy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EC (Active Comparator): Cyclophosphamide,600 mg/m2 q3wk and Epirubicin,90 mg/m2 q3wk
  Interventions: Drug: Epirubicin+Cyclophosphamide
- LC (Experimental): liposomal doxorubicin, 37.5 mg/m2 q3wk, and Cyclophosphamide,600 mg/m2 q3wk
  Interventions: Drug: liposomal-doxorubicin+Cyclophosphamide

INTERVENTIONS:
Drug: Epirubicin+Cyclophosphamide — Cyclophosphamide 600 mg/m2 infusion followed by epirubicin 90 mg/m2 infusion on Day 1 in each 21-day treatment cycle. Treatment will be repeated for 4 cycles in the EC arm.
  Arms: EC
Drug: liposomal-doxorubicin+Cyclophosphamide — Cyclophosphamide 600 mg/m2 infusion followed by pegylated liposomal-doxorubicin 37.5mg/m2 infusion on Day 1 in each 21-day treatment cycle. Treatment will be repeated for 5 cycles in the LC arm.
  Arms: LC

SUMMARY:
Primary objective:

* To evaluate the disease-free survival (DFS) in the two randomized arms after therapy with LC vs. EC in chemo-naive Her2-patients with stage I or II breast cancer

Secondary objectives:

* To assess the overall survival (OS)
* To establish the safety profile by assessing the toxicities and tolerability
* To assess the quality of life (QoL)
* To evaluate survival correlation with biomarkers expression.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed invasive, but non-inflammatory, breast adenocarcinoma with stage I or II (if N0, T must be >1cm) disease
* Her2-negative on fluorescence in situ hybridization (FISH) study
* performance status of ECOG 0, 1
* female, age between 20 and 70 years
* life expectancy of at least one year
* ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Her2 3+ over-expression on immunohistochemistry (IHC), or Her2 amplification on fluorescence in situ hybridization (FISH) study
* previous or current systemic malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ, unless there has been a disease-free interval of at least 5 years
* Patients who have received prior chemotherapy
* inadequate hematological function defined as absolute neutrophil count (ANC)less than 1,500/mm3, and platelets less than 100,000/mm3
* inadequate hepatic function defined as: serum bilirubin greater than 1.5 times the upper limit of normal range (ULN) alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than 2.5 times the ULN
* inadequate renal function defined as serum creatinine greater than 1.5 times the ULN
* left ventricular ejection fraction (LVEF) < 50% confirmed by multiple-gated acquisition (MUGA) scan or echocardiogram
* concomitant illness that might be aggregated by chemotherapy or interfere study assessment. For examples, active, non- controlled infection (such as hepatitis B and hepatitis C, HIV, infectious tuberculosis) or other active, non-controlled disease such as congestive heart failure, ischemic heart disease, uncontrolled hypertension or arrhythmia, unstable diabetes mellitus, and active peptic ulcer
* patients who are presence of liver cirrhosis or are HBV/HCV carrier
* participation in another clinical trial with any investigational drug within 30 days prior to entry
* pregnant or breast feeding women
* fertile women of child-bearing potential unless using a reliable and appropriate contraceptive method throughout the treatment period and for three months following cessation of treatment

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2010-06; Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  To evaluate the disease-free survival (DFS) in the two randomized arms after therapy with LC vs. EC in chemo-naive Her2-patients with stage I or II breast cancer

SECONDARY OUTCOMES:
Overall survival | 5 years
Quality of life | Baseline and every 3 weeks during therapy
Safety profiles | 5 years
  Incidence and severity of adverse event (neutropenia, palmar-plantar erythrodysesthesia, cardiac function, and secondary leukemia) by assessing the toxicities and tolerability
Survival correlation with biomarkers expression | At approximately of 5 years maximum FU

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Feng Hou, MD, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (9):
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang-Gung Memorial Hospital, Linkou, Linkou District
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei